CLINICAL TRIAL: NCT03007719
Title: Functional Imaging of T-Cell Activation With [18F]F-AraG in Urothelial Carcinoma Patients Receiving Neoadjuvant Therapy or Patients With Cancer Receiving Standard of Care Anti-PD-1/L1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Lawrence Fong (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Fong, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16709; NCI-2017-01323 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Neoadjuvant (Experimental): Patients with localized bladder cancer who are eligible for the UCSF phase 2 clinical trial of neoadjuvant atezolizumab before definitive surgery (NCT02451423) (Cohort 1). For the neoadjuvant cohort, study participants will undergo whole body PET/MR imaging with [18F]F-AraG within 7 days of initiating atezolizumab and within 7 days before surgery. Approximately 12 patients will be enrolled.
  Interventions: Drug: Fluorine F 18 Ara-G; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging
- Cohort 2: Standard of Care (SOC) (Experimental): Patients with any cancer type who are planned to initiate standard of care (SOC) anti-PD-1 or anti-PD-L1 treatment (Cohort 2). For the SOC cohort, study participants will undergo whole body PET/MR imaging with [18F]F-AraG within 7 days of initiating Cycle 1 anti-PD-1 or anti-PD-L1, and between Cycle 1 Day 15 (C1D15) and Cycle 2 Day 7 (C2D7) anti-PD-1 or anti-PD-L1. Approximately 19 patients will be enrolled.
  Interventions: Drug: Fluorine F 18 Ara-G; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Fluorine F 18 Ara-G — Given IV
  Other Names: 2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine; VisAcT
Procedure: Positron Emission Tomography — Undergo PET/MR imaging
  Other Names: PET; PET Scan
Procedure: Magnetic Resonance Imaging — Undergo PET/MR imaging
  Other Names: MRI

SUMMARY:
This phase II trial studies how well fluorine F 18 Ara-G positron emission tomography (PET)/magnetic resonance (MR) imaging works in measuring clinical response to atezolizumab or patients with cancer receiving standard of care Anti-PD-1/L1. Diagnostic procedures, such as fluorine F 18 Ara-G PET/MR imaging, may help measure a patient's response to standard of care atezolizumab or Anti-PD-1/L1 treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the change in fluorine F 18 Ara-G ([18F]F-AraG) uptake in primary and/or metastatic tumor(s) on whole-body [18F]F-AraG PET/MR imaging associated with neoadjuvant atezolizumab and standard of care (SOC) anti-PD-1 or anti-PD-L1 treatment.

SECONDARY OBJECTIVES:

I. To correlate change in [18F]F-AraG uptake within the primary tumor with clinical and pathologic response in patients treated with neoadjuvant atezolizumab. (Cohort 1) II. To assess [18F]F-AraG uptake in lymphoid organs before and after anti-PD-1 or anti-PD-L1 treatment. (Cohort 1 and 2)

OUTLINE: Patients are assigned to 1 or 2 cohorts.

COHORT I (NEOADJUVANT COHORT): Patients receive fluorine F 18 Ara-G intravenously (IV) and undergo PET/MR imaging over 1.5-3 hours within 7 days of starting standard of care atezolizumab and within 7 days before surgery.

COHORT II (SOC COHORT): Patients receive fluorine F 18 Ara-G IV and undergo PET/MR imaging over 1.5-3 hours within 7 days of initiating course 1 of anti-PD-1 or anti-PD-L1 therapy and between day 15 of course 1 and day 7 of course 2 of anti-PD-1 or anti-PD-L1 treatment.

After completion of study, patients are followed up at days 2 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented cancer to which anti-PD1 or anti-PDL1 are approved therapies
* Eligible for with plan to undergo neoadjuvant treatment with atezolizumab followed by surgery as part of a companion study (NCT02451423), or planned to undergo treatment with anti-PD-1 or anti-PD-L1 per standard of care
* Must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 regardless of disease stage (e.g. localized, locally advanced, or metastatic)
* In female patients, negative pregnancy test with no plans to become pregnant during the duration of the study
* Able to provide informed consent and follow the study guidelines
* Archival tumor tissue from biopsy or resection will be required for all patients; archival tissue should be of good quality based on total and viable tumor contents; fine needle aspiration, brushing, and cytologic cell pellets are not acceptable

Exclusion Criteria:

* History of prior treatment with immune checkpoint antibodies (e.g. anti-PD1, anti-PDL1, anti-CTLA4 antibody) or co-stimulatory agonist antibodies (e.g. anti-41BB, anti-OX40)

  * Prior intravesical treatment with Bacillus Calmette-Guerin (BCG) is allowed; however, the last dose must be at least 6 weeks from time of enrollment and patients must have documented progressive disease at least 6 weeks from completion of last BCG
* Diagnosis of immunodeficiency including history of human immunodeficiency virus (HIV)
* Receiving systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to first injection of [18F]F-AraG

  * Topical and inhaled corticosteroids are allowed
* Prior allogeneic stem cell or solid organ transplant
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Biopsy or resection of the primary tumor within 14 days the first injection of [18F]F-AraG
* Contraindication to magnetic resonance (MRI) imaging, as determined through review of the University of California, San Francisco (UCSF) MRI screening form by study investigator
* Evidence of active infection within 14 days of study enrollment
* Female patients who are pregnant or breastfeeding
* Inability to receive furosemide (Lasix) in the opinion of the treating investigator
* Patients that plan to receive off-label use of anti-PD1 or anti-PDL1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was closed due to low accrual. Only 4 patients were enrolled to this protocol and all were assigned to cohort 2
Groups:
- Cohort 1: Neoadjuvant: Patients with localized bladder cancer who are eligible for the University of California, San Francisco (UCSF) phase 2 clinical trial of neoadjuvant atezolizumab before definitive surgery (NCT02451423) (Cohort 1).
- Cohort 2: Standard of Care (SOC): Patients with any cancer type who are planned to initiate standard of care (SOC) anti-PD-1 or anti-PD-L1 treatment (Cohort 2).
Period: Overall Study
Arm/Group | Cohort 1: Neoadjuvant | Cohort 2: Standard of Care (SOC)
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only four participants were consented and enrolled to this protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Neoadjuvant | Cohort 2: Standard of Care (SOC) | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Customized [Count of Participants; unit: Participants]
  60-69 |  | 1 | 1
  70-79 |  | 2 | 2
  80-89 |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change Between Pre-treatment and Post-treatment SUVmax (Standardized Uptake Values) in the Primary and/or Metastatic Tumor(s) on Whole-body [18F]F-AraG Positron Emission Tomography/Magnetic Resonance (PET/MR) Imaging by Study Cohort.
Description: The nonparametric paired Wilcoxon Signed-rank test will be used to assess differences in SUVmax before and after treatment. The log2 ratio of post-treatment versus baseline SUVmax within the tumor and lymphoid tissues will also be calculated
Time Frame: Up to 2 weeks
Population: SUVmax data not collected
Arm/Group | Cohort 1: Neoadjuvant | Cohort 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Change in SUVmax of the Primary Tumor in Patients Who Achieve Pathologic Downstaging or Clinical Response and Those Without Pathologic or Clinical Response at Time of Surgery in Patients Receiving Neoadjuvant Atezolizumab (Cohort 1)
Description: To correlate change in SUVmax to clinical and/or pathologic response, patients will be divided into two groups: those who achieved clinical response and/or pathologic downs-staging, and those who did not. The median and interquartile range of change in SUVmax from baseline to pre-surgery in the different groups will be descriptively reported. For Cohort 1, clinical response will be determined by abdominal imaging performed <30 days after the last dose of atezolizumab prior to cystectomy compared to baseline pre-treatment imaging using RECIST v1.1 criteria, as specified in the companion treatment protocol. For Cohort 1, pathologic response will be determined by evidence of down-staging (e.g. from muscle invasive to non-muscle invasive, or complete pathologic response) at the time of cystectomy.
Time Frame: Up to 6 weeks
Population: SUVmax data not collected
Arm/Group | Cohort 1: Neoadjuvant
Number analyzed (Participants) | 0

3. Secondary Outcome: Change Between Pre-treatment and Post-treatment SUVmax in Lymphoid Organs on Whole-body [18F]F-AraG PET/MR Imaging (Cohort 1 and 2)
Time Frame: Up to 8 days
Population: SUVmax data not collected
Arm/Group | Cohort 1: Neoadjuvant | Cohort 2: Standard of Care (SOC)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were evaluated one day and one week via telephone visit after each radiopharmaceutical injection for safety follow-up, up to 6 weeks.
Description: No patients were enrolled in Cohort 1. All patients who receive any dose of [18F]F-AraG were analyzed for safety, all adverse events were recorded. Patients removed from study for unacceptable treatment related adverse event(s) were followed until resolution or stabilization of all treatment related adverse events (AE) to Grade 0-1.
Groups:
- Cohort 2: Standard of Care (SOC): Patients with any cancer type who are planned to initiate standard of care (SOC) anti-PD-1 or anti-PD-L1 treatment.
Arm/Group | Cohort 2: Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2: Standard of Care (SOC) (N=4)
Hematuria (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated due to low accrual. Only four participants were accrued to Cohort 2 (SOC) for this protocol. No patients were enrolled for cohort 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT03007719/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03007719/Prot_SAP_001.pdf